CLINICAL TRIAL: NCT05619289
Title: Immune Mechanisms of Vitamin D in a Randomized Controlled Trial to Reduce Chronic Pain After Burn
Brief Title: Immune Mechanisms of Vitamin D to Reduce Chronic Pain After Burn
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22-1310; K23AT011389-01A1 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Burn Injury; Chronic Pain
MeSH Terms: conditions — Burns; Chronic Pain | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D2 (Ergocalciferol) (Active Comparator): One time, oral dose of Vitamin D2 administered via 6 50,000 IU Ergocalciferol capsules. Capsules will be encapsulated and masked to be indistinguishable from placebo.
  Interventions: Drug: Ergocalciferol
- Placebo (Placebo Comparator): One time, oral dose of 6 placebo capsules filled with inert powder and encapsulated and masked to be indistinguishable from active comparator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ergocalciferol — One-time, oral dose of 300,000 IU of Ergocalciferol administered via 6 capsules.
  Other Names: Vitamin D2, Calciferol, Drisdol
  Arms: Vitamin D2 (Ergocalciferol)
Drug: Placebo — One-time, oral dose of 6 inert capsules matched to the active comparator
  Arms: Placebo

SUMMARY:
The goal of this pilot clinical trial is to learn whether vitamin D is able to prevent chronic pain following burn injury and to determine what biological mechanisms are engaged by Vitamin D following burn injury. The main question[s] it aims to answer are:

* Is the clinical trial protocol feasible?
* Is Vitamin D administration following burn injury safe?
* How does vitamin D cause changes in the immune system in the aftermath of burn injury?

Following informed consent, participants will be asked to:

* Take 6 capsules by mouth one time following burn injury (Vitamin D or Placebo)
* Provide a blood sample at baseline and 6 weeks following injury
* Fill out surveys daily while in the hospital, weekly through 6 weeks, and at 3 months and 6 months.

Researchers will compare Vitamin D and placebo groups to see if there are differences in adverse effects (side effects), chronic pain, and profiles of immune cells from collected blood samples.

ELIGIBILITY:
Inclusion Criteria

* ≥ 18 years and ≤ 70 years of age
* MThBI severe enough to warrant admission to Burn Surgery Service (NOTE: surgery may or may not be indicated)
* Admission and subsequent enrollment occurs within 1 week of MThBI
* Patients experience a thermal burn injury, not an electrical or chemical burn.
* Has a smartphone with continuous service >1 year
* Alert and oriented
* Willing to take study medication (6 capsules of Vitamin D or placebo)
* Point of care Vitamin D level <100 ng/mL
* Able to speak and read English
* Burn survivors with acute pain severity ≥ 7/10 on the Numeric Rating Scale (initial pain severity reported by patient on screening)
* Total Body surface area burned <30%

Exclusion Criteria

* Substantial comorbid injury (e.g. long bone fracture)
* Pregnancy/Breastfeeding
* Prisoner status
* Active psychosis, suicidal ideation, or homicidal ideation
* Requires an emergency/bedside escharotomy or fasciotomy for the treatment of burn injury.
* Known Child-Pugh liver disease severity classification B or C.
* Known chronic kidney disease stage 4 or higher (GFR≤29).
* No other history or condition that would, in the investigator's judgment, indicate that the patient would very likely be non-compliant with the study or unsuitable for the study (e.g. might interfere with the study, confound interpretation, or endanger patient).
* Intubated and sedated at time of enrollment.
* Hypersensitivity to Vitamin D3, ergocalciferol, calcitriol, alfacalcidol, calcipotriol
* Known hypercalcemia (based on routine admission laboratory assessment).
* Sarcoidosis
* Hyperphosphatemia (based on routine admission laboratory assessment)
* Taking Vitamin D supplements in excess of 800 IU daily.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Follow-up rate 6 weeks following burn injury | 6 weeks
  The proportion of patients who are able to follow-up at 6 weeks and complete a questionnaire will be calculated. To meet the primary outcome, follow-up will be >80% at 6 weeks.

SECONDARY OUTCOMES:
25-hydroxyvitamin D concentration 6 weeks after Vitamin D2 treatment | Baseline, 6 weeks
  Measure the ability of Vitamin D administration to generate sustained increases in whole-blood Vitamin D concentrations (nanograms per deciliter (ng/dl), between baseline and 6 weeks. 25-hydroxyvitamin D concentration will be determined by performing mass spectroscopy on blood spot cards collected at enrollment and at 6 weeks to determine circulating Vitamin D concentration in ng/dl. Mean concentration change from baseline and 6 weeks will be reported for participants in the placebo and intervention group.
Safety of Vitamin D2 administration in aftermath of burn injury | 6 weeks
  To assess safety, adverse events will be tracked through surveys during the 6 weeks after treatment to assess side effects and safety profile of Vitamin D. Adverse Events will be reported using Common Terminology Criteria for Adverse Events (CTCAE). Events will be graded in severity with grade 3 representing severe, grade 4 representing life-threatening, and grade 5 representing death. Relatedness will be categorized as unrelated, unlikely, possible, probable, definite. For this safety measure, we will report the number of grade 3 or higher severity and probable or higher relatedness in the placebo and intervention groups.
By Group Efficacy Estimates Over Year Following Thermal Burn Injury | Baseline, 1 week, 2 week, 3 week, 4 week, 5 week, and 6 weeks, 3 months, 6 months
  Preliminary estimates of efficacy (95% confidence intervals) will be obtained via repeated measures analysis of pain severity over the 1 year following injury using mixed effects models. Pain will be assessed using a 0-10 numeric rating scale with 0 indicating no pain and 10 indicating pain as severe as you can imagine. Higher scores represent worse outcome. These values (collected in identical fashion over 6 months following burn injury) will be entered into a linear mixed model, and overall effect estimates (beta coefficients) among groups will be determined. Unadjusted values will be reported as well as after for adjusting for baseline psychosocial factors (pain catastrophizing, anxiety, depression, stress, perceived social support), sociodemographic factors (age, sex, ethnicity, income, education attainment), and wound healing-related factors. This will be reported over the study period.
Opioid cessation | 6 months
  Opioid cessation will be defined as the date in which opioids are discontinued for three consecutive days. Median time (days) to opioid cessation will be reported for the treatment and placebo groups.
Neuropathic pain quality | 6 months
  Use NIH Patient-Reported Outcomes Measurement Information Systems (PROMIS) Neuropathic pain quality to assesses to what degree (from"not at all" to " very much") the respondent's pain shows qualities typical of neuropathic pain in the past 7 days using a 1-5 scale, where 1 indicates "not at all" and 5 indicates "very much." The total scale represented on a scale from 5-25 with 25 representing the highest level of neuropathic pain. This total scale value will be reported for placebo and intervention groups 6 months following treatment.
Pain Interference | 6 months
  Use NIH PROMIS Pain interference to determine the extent to which pain interferes with life function. Participants are assessed the degree to which pain interferes with life function across 8 domains. The participants rates interference on a scale of 1 to 5 with 1 representing no interference and 5 representing the maximum interference. The total scale represented on a scale of 8-40 with 40 representing the most interference. Raw scores will be converted to a T score with standard error represented in the derived measure look-up table provided by the NIH PROMIS website. T-scores will be reported for the placebo and intervention groups 6 months following treatment.
Widespread pain severity | 6 months
  Regional Pain Scale (RPS) will be used to assesses pain presence (yes=1, no=0), and severity if present using a 0-10 numeric rating scale. 0-10 scale where 0 indicates no pain and 10 is the worst pain imaginable, for each location of the body (right arm, right, leg, trunk, etc). The mean number of body regions reported as painful (numeric rating scale greater than or equal to 4) will be reported for placebo and intervention groups.
Nociceptive quality | 6 months
  Nociceptive quality of pain will be determined with the NIH PROMIS Nociceptive Pain Quality. Assesses to what degree (from"not at all" to " very much") the respondent's pain shows qualities typical of nociceptive pain in the past 7 days using a 1-5 scale, where 1 indicates "not at all" and 5 indicates "very much." The total scale represented on a scale from 5-25 with 25 representing the highest level of nociceptive pain. Mean total score will be reported for placebo and intervention groups.

OTHER OUTCOMES:
Inflammatory immune cells populations assessed with mass cytometry | 6 weeks
  Use a custom antibody panel to assess immune cell frequency, and Toll-like receptor 4 (TLR4) activation with phosphorylated NFkB (p-NFkB) as a readout for TLR4 activation). The proportion of immune cells will be determined. Immune cell frequencies multiple parallel mediation model to determine whether immune cells mediate Vitamin D treatment effects. This is an exploratory analysis. Mean proportions of monocytes, cluster of differentiation (CD) 4 T-cells, CD 8 T-cells, neutrophils, mast cells, natural killer-cells will be reported for placebo and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mauck, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University Of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared on request provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 12 and continuing for 36 months after publication
Access Criteria: Approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.